CLINICAL TRIAL: NCT01384890
Title: Feasibility of Volumetric Modulated Arc Therapy and Cone-Beam Computed Tomography for Head and Neck Carinomas: Analysis of Clinical Throughput and Patient Reported Outcomes.
Brief Title: Feasibility of VMAT and CBCT for Head and Neck Carcinomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Principal Investigator, Jonn Wu, Dr. Jonn Wu, British Columbia Cancer Agency
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VMAT, CBCT for H&N ca
Record Dates: First submitted 2011-06-28; First posted 2011-06-29 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2013-02

CONDITIONS: Head and Neck Carcinoma
MeSH Terms: interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- VMAT with CBCT (Experimental): Volumetric modulated arc therapy (VMAT) with cone-beam computed tomography position (CBCT) verification
  Interventions: Radiation: VMAT with CBCT
- VMAT with kV-ray (Active Comparator): Volumetric modulation arc therapy (VMAT) with kV-ray position verification
  Interventions: Radiation: VMAT with kV-ray

INTERVENTIONS:
Radiation: VMAT with CBCT — volumetric modulated arc therapy (VMAT) with cone-beam computed tomography (CBCT) position verification
  Arms: VMAT with CBCT
Radiation: VMAT with kV-ray — Volumetric modulated arc therapy (VMAT) with kV-ray position verification
  Arms: VMAT with kV-ray

SUMMARY:
This will be a prospective longitudinal study describing clinical throughput metrics and patient reported quality of life outcome measures for patients undergoing Volumetric modulated arc therapy (VMAT) with and without Cone-beam computed tomography (CBCT) for head and neck carcinoma at the British Columbia Cancer Agency.

1. VMAT for the treatment of patients with HNC will provide opportunities for image-guided radiotherapy using CBCT online correction to reduce systematic and random error.
2. Analysis of patient reported quality of life outcomes during VMAT, with and without CBCT acquisition, will be hypothesis generating.

ELIGIBILITY:
Inclusion Criteria:

* age greater than 18 years
* undergoing radical radiation therapy for head and neck carcinoma at the BC Cancer Agency

Exclusion Criteria:

* treatment being offered is not for curative intent
* patient has received previous radiation for head and neck cancer
* patient has systemic lupus erythematosis or scleroderma
* patients has other autoimmune connective tissue disorders

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-07; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Clinical efficiency for volumetric modulated arc therapy (VMAT) delivery | After patient treated
  Prospective work-flow metrics describing clinical efficiency for volumetric modulated arc therapy (VMAT) delivery with and without cone-beam computed tomography (CBCT) acquisition at the BCCA, generated from time requirements for treatment verification and delivery. The time spent by the patients at each stage of radiation therapy delivery will be recorded, including; time in radiation bunker, time in immobilization frame, kV or CBCT acquisition and online correction time, and beam on time
Position verification | After patient treated
  Summary description of position verification and online corrections for volumetric modulated arch therapy (VMAT) delivery with and without cone-beam computed tomography (CBCT)

SECONDARY OUTCOMES:
Quality of life | No time frame (ongoing)
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire for Head and Neck Cancer (EORTC QLQ - HN35) (23) (see Appendix V) and State Trait Anxiety Index (STAI)

CONTACTS AND LOCATIONS:
Overall Officials: Jonn Wu, MD, Principal Investigator — British Columbia Cancer Agency
Locations (1):
- BC Cancer Agency - Vancouver Centre, Vancouver, British Columbia, Canada